CLINICAL TRIAL: NCT02347254
Title: Feasibility Trial Evaluating the Safety and Efficacy of ExAblate Transcranial Magnetic Resonance Guided Focused Ultrasound (MRgFUS) for Unilateral Pallidotomy for the Treatment of L-Dopa Induced Dyskinesia (LID) of Parkinson's Disease.
Brief Title: ExAblate Transcranial MRgFUS for Unilateral Pallidotomy for the Treatment of Parkinson's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD004; 222434 (Other: Canada: Health Canada)
Record Dates: First submitted 2015-01-12; First posted 2015-01-27 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transcranial ExAblate (Experimental): Transcranial ExAblate MRgFUS
  Interventions: Device: Transcranial ExAblate

INTERVENTIONS:
Device: Transcranial ExAblate — Transcranial ExAblate MRgFUS
  Other Names: ExAblate; TcMRgFUS

SUMMARY:
The proposed study is to evaluate the safety and initial effectiveness of the ExAblate Transcranial MRgFUS) treatment of patients with L-dopa induced dyskinesia of Parkinson's disease (LID PD).

Safety:

To evaluate the incidence and severity of adverse events associated with ExAblate Transcranial 4000 MRgFUS treatment of dyskinesia of Parkinson's disease.

Effectiveness:

To determine the level of effectiveness of the ExAblate Transcranial MRgFUS treatment of LID in PD patients. Efficacy will be determined utilizing clinical rating scales for dyskinesia (UPDRS-IV and the Unified Dyskinesia Rating Scale) from examinations at Baseline, 3-Months and 12-Months post-ExAblate treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, between 18 and 80 years, inclusive.
* Patients who are able and willing to give consent and able to attend all study visits.
* Able to communicate sensations during the ExAblate MRgFUS treatment
* Stable doses of all medications for 30 days prior to study entry and for the duration of the study.
* Inclusion and exclusion criteria have been agreed upon by two members of the medical team.

Exclusion Criteria:

* Patients with unstable cardiac status including:
* Unstable angina pectoris on medication
* Patients with documented myocardial infarction within six months of protocol entry
* Congestive heart failure requiring medication (other than diuretic)
* Patients on anti-arrhythmic drugs
* Severe hypertension (diastolic BP > 100 on medication)
* Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
* Known intolerance or allergies to the MRI contrast agent (e.g. Gadolinium or Magnevist) including advanced kidney disease
* Severely impaired renal function (estimated glomerular filtration rate < 30ml/min/1.73 m2) or receiving dialysis
* History of abnormal bleeding and/or coagulopathy
* Cerebrovascular disease (multiple CVA or CVA within 6 months)
* Symptoms and signs of increased intracranial pressure (e.g. headache, nausea, vomiting, lethargy, and papilledema)
* Active or suspected acute or chronic uncontrolled infection
* History of intracranial hemorrhage
* Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
* Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment
* Are participating or have participated in another clinical trial in the last 30 days
* Patients unable to communicate with the investigator and staff.
* Presence of any other neurodegenerative disease like parkinson-plus syndromes suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, dementia with Lewy bodies, and Alzheimer's disease.
* Presence of significant cognitive impairment as determined with a score <= 24 on the Mini Mental Status Examination (MMSE)
* Patients with a history of seizures within the past year
* Patients with psychiatric illness that are not well controlled. Any presence of psychosis will be excluded. Patients with mood disorders including depression will be excluded if they have exhibited symptoms within 6 months while on medication. Patients who have been treated with transcranial magnetic stimulation or ECT will be excluded.
* Patients with risk factors for intraoperative or postoperative bleeding (platelet count less than 100,000 per cubic millimeter) or a documented coagulopathy
* Patients with brain tumors
* Any illness that in the investigator's opinion preclude participation in this study.
* Pregnancy or lactation.
* Patient is unable to provide their own consent for any reason.
* Legal incapacity or limited legal capacity.
* Patients who have had deep brain stimulation or a prior stereotactic ablation of the basal ganglia
* History of immunocompromise, including patient who is HIV positive
* Known life-threatening systemic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2014-09; Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of Device and Procedure related adverse events | At the time of ExAblate trascranial procedure
  To evaluate the incidence and severity of adverse events associated with ExAblate Transcranial 4000 MRgFUS treatment of dyskinesia of Parkinson's disease.

SECONDARY OUTCOMES:
Severity of Device and Procedure related adverse events | At the time of ExAblate trascranial procedure
  To evaluate the incidence and severity of adverse events associated with ExAblate Transcranial 4000 MRgFUS treatment of dyskinesia of Parkinson's disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada